CLINICAL TRIAL: NCT06801340
Title: Assessment of Metabolic Complications in Patients With Adrenal Tumors Through Radiological Images
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RADIO-AT
Record Dates: First submitted 2024-12-30; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Adrenal Cancer
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study based on data already available at each Center. Pseudonymized CT images of each patient in DICOM format will be sent from each center to the Coordinating Center to perform radiomics analysis.

DETAILED DESCRIPTION:
Retrospective study based on data already available at each Center. Participating Centers will identify patients based on shared inclusion/exclusion criteria. Pseudonymized CT images of each patient in DICOM format will be sent from each center to the Coordinating Center to perform radiomics analysis. Images will be transferred via File Transfer Protocol while respecting the anonymity of enrolled patients. Images will be deposited in a dedicated study folder created by the AOUBO ICT Service. Images will be accessible only to the Investigator and Principal Investigator and/or their delegates via personalized credentials, which can be accessed only from IRCCS AOUBO computers and facilities. The folder to which the images will be transferred will be accessible only to the Principal Investigator and his/her Collaborators through customized private credentials usable only through IRCCS AOUBO networks, computers and facilities. Radiomics, which will be applied to existing CT images, will in no way affect the care pathway of patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with adrenal tumor who underwent adrenectomy surgery from 1-1-2000 to 30-5-2023, performed according to clinical necessity and indications of international guidelines,with availability of histologic diagnosis or adrenal tumor that did not undergo adrenectomy surgery with diagnosis of benignity confirmed by radiologic stability at 6-12 months after first finding(as indicated in guidelines)
* Availability of radiological images in DICOM format of abdominal CT scan in which the adrenal tumor is first described, obtained on the date of first evaluation at the participating center (necessarily before surgery for patients undergoing adrenectomy)
* Signature of informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the study will be enrolled at participating centers, selected from those who meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Radiomics-Derived Parameters for Differentiating Benign and Malignant Adrenal Masses | through study completion, an average of 1 year
  This measure will assess the diagnostic ability of specific radiomics-derived parameters, including texture analysis and intensity features, in identifying the nature (benign or malignant) of adrenal masses. The diagnostic performance will be evaluated through sensitivity, specificity.

SECONDARY OUTCOMES:
Association of Radiomics-Derived Parameters with Ki67 Values | through study completion, an average of 1 years
  This measure evaluates the correlation between radiomics-derived imaging parameters and Ki67 proliferation index values. Ki67 values will be assessed as a percentage using immunohistochemical staining, and the correlation will be expressed as a Pearson or Spearman correlation coefficient, depending on data distribution.
Association of Radiomics-Derived Parameters with Weiss' Anatomopathologic Score | through study completion, an average of 1 year
  This measure evaluates the correlation between radiomics-derived imaging parameters and the Weiss anatomopathologic score. The Weiss score will be determined based on pathological examination, and the association will be reported as a correlation coefficient.
Association of Radiomics-Derived Parameters with Occurrence of Distant Metastasis | through study completion, an average of 1 year
  This measure evaluates the relationship between radiomics-derived imaging parameters and the occurrence of distant metastases in patients with adrenal tumors. The occurrence of metastases will be reported as a binary outcome (presence or absence), and the association will be analyzed using logistic regression models or similar statistical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Di Dalmazi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No